CLINICAL TRIAL: NCT01447498
Title: Effect of a Systematic Screening for Risk-factors for Ulcer Bleeding Before Post-PCI Anti-thrombotic Treatment
Brief Title: Systematic Screening for Risk-factors for Ulcer Bleeding Before Anti-thrombotic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Danish Heart Foundation (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Berit Elin Søltoft Jensen, MD sub-investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Projekt ASA
Record Dates: First submitted 2011-09-26; First posted 2011-10-06 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Occlusion/Thrombosis; Peptic Ulcer Hemorrhage
MeSH Terms: conditions — Coronary Occlusion; Thrombosis; Peptic Ulcer Hemorrhage | interventions — Mass Screening; Risk Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention)
- Screening and risk assessment (Active Comparator)
  Interventions: Other: Screening for risk factors for ulcer bleeding

INTERVENTIONS:
Other: Screening for risk factors for ulcer bleeding — Following PCI the patients fill out a questionnaire to assess the risk factors for ulcer bleeding.We randomise between:
  1. screening and risk assessment
  2. control group
  All screened patients, who fulfil the criteria for having a moderate to high risk of ulcer bleeding will be sent written information about risk factors and the purpose of the PPI prophylaxis. They will be recommended PPI prophylaxis (Pantoprazole), as long as they are being treated with low-dose aspirin and clopidogrel.
  Patients in the screening group, who are already on PPI treatment is recommended to change to Pantoprazole.
  Definition of risk of ulcer bleeding: The table below will be used for screening. Patients scoring ≥ 2 points will receive PPI prophylaxis.
  points: Age: < 60: 0; 60-69: 1; 70-79: 2; >=80: 3 ___ Dyspepsia: 1 ___ Uncomplicated ulcer: 2 ___ Complicated ulcer 3 ___ NSAID 2 ___ Steroids 2 ___ SSRI 2 ___ Anticoagulant Tx 2 ___
  Arms: Screening and risk assessment

SUMMARY:
In a prospective randomised study design to investigate, if a systematic risk factor screening for bleeding ulcer in patients, who following percutaneous coronary intervention (PCI) commence a one year combination treatment with low dose aspirin and clopidogrel, followed by prophylactic treatment with a proton pump inhibitor (PPI) in case of increased risk, can reduce the risk of bleeding ulcer. Based on the recently raised suspicion that PPI's, possibly except pantoprazole, reduce the effect of ADP-receptor inhibitors, pantoprazole has been chosen as prophylaxis in the screening group, and analyses will be done to ascertain whether PPI treatment increases the risk of coronary events. Further analyses will be made to see whether PPI prophylaxis in high risk patients can increase compliance with the antithrombotic treatment through a reduction of side effects, thereby reducing the risk of myocardial infarction in particular stent thrombosis. The study population will be analyzed further to identify the patients, who will benefit the most from PPI prophylaxis Hypothesis: screening heart patients for risk factors for bleeding ulcer and subsequently treating high risk patients with PPI can reduce the incidence of bleeding ulcer and increase compliance with the antithrombotic treatment; thereby possibly reducing the risk of coronary events and improving survival. Initial a description of the prevalence of risk factors will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients who has had a PCI with stenting or balloon dilatation in the cardiology department at Odense University Hospital, Århus University Hospital and Ålborg Sygehus, where subsequent treatment with low-dose aspiring and clopidogrel or another thienopyridine is planned for one year.

Exclusion Criteria:

* previous PCI with stenting or balloon dilatation
* treatment with clopidogrel prior to PCI
* lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2024 (Actual)
Dates: Start 2011-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Admission for ulcer bleeding or haemorrhagic gastritis | 1 year
  Efficacy of a systematic screening for risk factors for ulcer bleeding in patients, who after percutaneous coronary intervention (PCI), is treated with antithrombotic medicine

SECONDARY OUTCOMES:
Compliance with antithrombotic medicine | 1 year
  Does prophylactic treatment with proton pump inhibitor increase the compliance with antithrombotic medicine and thereby decrease the risk of new cardiac event.
Identification of patients with benefit of proton pump inhibitor prophylaxis | 1 year
  Analysis of risk factors is planned in order to define which patients have the greatest benefit of PPI prophylaxis when receiving antithrombotic treatment.
Gastrointestinal bleeding | 1 Year
  Admission to hospital for not endoscopic verified upper gastrointestinal bleeding.
Uncomplicated ulcers | 1 year
  Development of uncomplicated ulcers
Death | 1 Year
  Registration of cause of death
Acute coronary syndrome | 1 Year
  Re-admission for acute coronary syndrome, including stent occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark